CLINICAL TRIAL: NCT06274489
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of the NOX1/4 Inhibitor Setanaxib in Patients With Alport Syndrome
Brief Title: A Study to Evaluate Setanaxib in Patients With Alport Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSN000500
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Alport Syndrome
MeSH Terms: conditions — Nephritis, Hereditary | interventions — setanaxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Setanaxib (Experimental): Patients will receive the following setanaxib doses according to age at the time of consent/assent:
  * For patients aged 12 to 17 years 1200 mg/day: 2 tablets in the morning (800 mg) and 1 tablet in the evening (400 mg)
  * For patients aged ≥18 years 1600 mg/day: 2 tablets in the morning (800 mg) and 2 tablets in the evening (800 mg)
  Interventions: Drug: Setanaxib
- Setanaxib placebo (Placebo Comparator): Matching placebo will be provided.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Setanaxib — Setanaxib (formerly GKT137831) is a first-in-class inhibitor of the human protein NADPH NOX1/4. It is a low molecular weight organic molecule and a member of the pyrazolopyridine dione chemical class.
  Arms: Setanaxib
Drug: Placebo — Matching film-coated placebo tablets, containing only excipients
  Arms: Setanaxib placebo

SUMMARY:
The purpose of the study is to learn about the safety and tolerability of setanaxib in subjects with Alport syndrome, when added to their standard of care treatment. The study will assess how safe setanaxib is when compared to placebo. Study participants will be asked if they are experiencing any side effects at each study visit. In addition, tests in blood, urine and other examinations will be used to look at the safety of setanaxib. The study will also measure how well setanaxib works in comparison to a placebo, by measuring urine protein and certain markers in the blood and urine. The concentration of setanaxib in the blood will also be measured throughout the course of the study.

Setanaxib is planned for use together with the current standard of care to hopefully provide additional therapeutic benefits by preserving kidney function.

The study will be conducted at multiple research sites in the UK, Spain, and Czech Republic. Eligible participants will be randomly assigned to receive either setanaxib or placebo. Setanaxib dose level will depend on age and all participants will receive their standard of care in addition to setanaxib or placebo. The study consists of a Screening period of up to 4 weeks, a 24-week Treatment period and a 4- week Follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 12 to 50 years inclusive, at the time of informed consent/assent. For sites in the European Union: Male or female patients aged 18 to 50 years, inclusive, at the time of informed consent;
2. Diagnosis of Alport syndrome by genetic testing (documented mutation in a gene associated with Alport syndrome [ie, COL4A3, COL4A4, or COL4A5]); Patients with a variant of uncertain significance should not be included in the study;

   Note: Genetic test results are to be available prior to initiating other Screening procedures. In cases where genetic testing results are not available but the patient is likely to fulfill the other inclusion and exclusion criteria and has provided consent/assent, a sample for genetic testing should be processed locally and the Screening Period duration can be prolonged with the time it takes to receive the genetic test results. All other Screening assessments must be completed within 4 weeks (± 7 days) prior to randomization.
3. Weight ≥40 kg;
4. Willing and able to give informed consent (and assent, where applicable), in accordance with local age requirements, and to comply with the requirements of the study;
5. Female patients of childbearing potential must use a highly effective method of contraception to prevent pregnancy for ≥4 weeks before randomization and must agree to continue strict contraception (as specified in 5c) up to 90 days after the last dose of investigational medicinal product (IMP);

   1. For the purposes of this study, women of childbearing potential (WOCBP) are defined as "fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy";
   2. Postmenopausal state is defined as no menses for 12 months without an alternative medical cause. In female patients who are not using hormonal contraception or hormonal replacement therapy but with suspected menopause and less than 12 months of amenorrhea, a high follicle-stimulating hormone level in the postmenopausal range will be required at Screening to confirm a postmenopausal state; and
   3. Highly effective contraception is defined as methods that can achieve a failure rate of less than 1% per year when used consistently and correctly. These methods include the following:

      * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal);
      * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable);
      * Intrauterine device;
      * Intrauterine hormone-releasing system;
      * Bilateral tubal occlusion;
      * Vasectomized partner; and
      * Sexual abstinence (refraining from heterosexual intercourse during the entire period of risk associated with the study treatments, ie, up to 90 days after the last dose of IMP). The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (calendar, symptothermal, or post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.
6. Female patients of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Visit 3 (after randomization and before dosing);
7. Male patients with female partners of childbearing potential must be willing to use a condom and require their partner to use a highly effective contraceptive method (as defined in the list in inclusion criterion 5c). Female condom and male condom should not be used together. This requirement begins at the time of informed consent/assent and ends 90 days after receiving the last dose of IMP;
8. Male patients must be willing not to donate sperm and female study patients must be willing not to donate eggs from baseline until 90 days after the last dose of IMP;
9. Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 at Study Visit 1 or 2, calculated at the central laboratory using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula for patients ≥18 years of age and the revised bedside Schwartz formula for patients 12 to 17 years of age;
10. Proteinuria (urine protein to creatinine ratio [UPCR] ≥90 mg/mmol [0.8 g/g]) at 2 consecutive measurements (24-hour urine sampling), separated by at least 2 weeks and calculated by the central laboratory;
11. Receiving maximum allowed dose or maximum-tolerated daily dose of an angiotensin-converting enzyme inhibitor (ACEi) and/or angiotensin II type I receptor blocker (ARB) that has been stable for at least 8 weeks prior to consent/assent; and Note: A stable dose is defined as a dose within 25% of the dose at randomization. Note: Patients with proven intolerance to ACEi and ARB are allowed in the study.

    Note: Sodium/glucose co-transporter 2 inhibitors are allowed provided they have been given at the same dose for at least 8 weeks prior to Screening and are given at the same dose during the study.
12. Systolic and diastolic blood pressure ≤95th percentile, based on the patient's age and height for patients 12 to 17 years of age or with ≤130 mmHg systolic blood pressure and ≤80 mmHg diastolic blood pressure for patients ≥18 years of age. Note: At least 1 blood pressure measurement during Screening (Study Visit 1 or 2) should be within these limits. Blood pressure will be measured after resting in the supine position for at least 5 minutes and will be measured 3 times with each measurement separated by at least 1 minute (the lowest value will be recorded on the electronic case report form).

Exclusion Criteria:

1. Has ongoing chronic hemodialysis or peritoneal dialysis;
2. Has a history of kidney transplant;
3. Has other causes of chronic kidney disease (CKD) (even if not yet on hemodialysis), including but not limited to other heritable disorders leading to CKD, diabetic nephropathy, hypertensive nephropathy, lupus nephritis, and immunoglobulin A nephropathy;
4. Has been treated with any investigational agent within 12 weeks of signing informed consent/assent or 5 half-lives of the investigational agent (if known), whichever is longer, or current enrollment in an interventional clinical study;
5. Has had prior treatment with setanaxib;
6. Has known malignancy that is progressing or requires active treatment, with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer that has undergone potentially curative therapy, or malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of study drug and of low potential risk for recurrence;
7. Positive urine drug screen (if not due to prescription use of a concomitant medication, as confirmed by the Investigator) at Screening. Patients on stable methadone or buprenorphine maintenance treatment for at least 6 months prior to Screening Visit 1 may be included in the study. Medicinal cannabis and cannabidiol products are not exclusionary and may be allowed if the prescription and diagnosis are reviewed and approved by the Investigator;
8. Has an active HIV infection or acute or chronic hepatitis B or C infection, confirmed at Screening;
9. Has had a surgery (eg, gastric bypass) or medical condition that might significantly affect absorption of medicines (as judged by the Investigator);
10. Has a positive pregnancy test at Study Visit 2 (Screening) and/or Study Visit 3 (Day 1) (WOCBP only) or is breastfeeding; Note: If a randomized patient has a positive pregnancy test at Study Visit 3 (Day 1), they will be considered a patient withdrawn for non-safety reasons.
11. Has evidence of any of the following cardiac conduction abnormalities at Screening or Day 1 (pre-dose): a QTcF interval >450 milliseconds for male patients or >470 milliseconds for female patients, or a PR interval ≥220 milliseconds; Note: Patients with a second or third degree atrioventricular block are to be excluded.
12. Has a history of aplastic anemia, or any current marked anemia, defined as hemoglobin <10.0 g/dL;
13. Has uncontrolled hypothyroidism. Patients with subclinical hypothyroidism may be included. Subclinical hypothyroidism is defined biochemically as a normal serum free thyroxine (T4) concentration in the presence of an elevated serum thyroid-stimulating hormone (TSH) concentration;
14. Has any laboratory abnormality or condition that, in the opinion of the Investigator, could interfere with or compromise a patient's treatment, assessment, or compliance with the Protocol and/or study procedures;
15. Has any other condition that, in the opinion of the Investigator, constitutes a risk or contraindication for the participation of the patient in the study, or that could interfere with the study objectives, conduct, or evaluation;
16. Uses medications known to be potent cytochrome P450 (CYP) 3A4 inhibitors (itraconazole, lopinavir/itonavir, telaprevir, clarithromycin, ritonavir, ketoconazole, indinavir/ritonavir, conivaptan, and voriconazole), potent CYP3A4 inducers (avasimibe, carbamazepine, enzalutamide, mitotane, nevirapine, phenobarbital, phenytoin, rifabutin, rifampicin, rifapentine, and St John's wort), or potent uridine 5'-diphospho-glucuronosyltransferase 1A9 inhibitors and inducers (mefenamic acid and rifampicin) within 21 days prior to study drug administration;
17. Has known psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring adverse events (AEs), or compromise the ability of the patient to give written informed consent/assent;
18. Has known hypersensitivity or intolerance to setanaxib or to any of its excipients;
19. Has a history of chronic liver disease (eg, primary biliary cholangitis, alcoholic liver disease, chronic viral hepatitis including hepatitis B and C, non-alcoholic fatty liver disease, and hemochromatosis);
20. Has plasma alanine aminotransferase and/or aspartate aminotransferase >3 x the upper limit of normal (ULN) at Study Visit 1 or 2 (Screening);
21. Has total bilirubin >2 x ULN at Study Visit 1 or 2 (Screening); or
22. Has international normalized ratio >1.2 at Study Visit 1 or 2 (Screening) (criterion not applicable for patients on anticoagulant therapy).

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Serious Adverse Events (SAEs) | From informed consent up to 30 days post-final dose
  Count and percentage of patients experiencing SAEs
Percentage of patients with treatment-emergent Adverse Events of Special Interest (AESIs) | From informed consent up to 30 days post-final dose
  Count and percentage of patients experiencing treatment-emergent AEISIs. CTCAE Grade ≥2 anemia will be considered an AESI. During the course of the study, additional AESIs may be identified by the Sponsor

SECONDARY OUTCOMES:
The ratio of urine protein to creatinine ratio (UPCR) analysed in 24-hour urine sample | At baseline and week 24
Percentage of patients with a 25% reduction in UPCR analysed in 24-hour urine sample | At baseline and week 24
  The proportions of patients achieving a 25% reduction in UPCR at 24 weeks from baseline in the setanaxib group will be compared to placebo group
The ratio of estimated glomerular filtration rate (eGFR) at 24 weeks compared to baseline. | At baseline and Week 24.
Pre-dose and post-dose plasma concentrations of setanaxib and GKT138184 measured as the area under the concentration-time curve over 24 hours at steady state (AUC0-24-ss) | within 90 minutes prior to dose and 0-, 1-, 2-, 3-, 4- and 6-hours post-dose at week 2; and prior to dose at weeks 12 and 24
Pre-dose and post-dose plasma concentrations of setanaxib and GKT138184 measured as the minimum plasma concentration at steady state (Cmin-ss) | within 90 minutes prior to dose and 0-, 1-, 2-, 3-, 4- and 6-hours post-dose at week 2; and prior to dose at weeks 12 and 24
Pre-dose and post-dose plasma concentrations of setanaxib and GKT138184 measured as the maximum plasma concentration at steady state (Cmax-ss) | within 90 minutes prior to dose and 0-, 1-, 2-, 3-, 4- and 6-hours post-dose at week 2; and prior to dose at weeks 12 and 24

OTHER OUTCOMES:
Percentage of patients with clinically significant changes in heart rate | From baseline by visit up to week 28 (study visit 9, Follow-Up)
  Clinically significant changes in heart rate from baseline by visit. Heart rate will be measured after resting in the supine position for at least 5 minutes and will be measured 3 times with each measurement separated by at least 1 minute (the lowest value will be recorded)
Percentage of patients with clinically significant changes blood pressure | From baseline by visit up to week 28 (study visit 9, Follow-Up)
  Clinically significant changes in blood pressure from baseline by visit. Systolic and diastolic blood pressure will be measured after resting in the supine position for at least 5 minutes and will be measured 3 times with each measurement separated by at least 1 minute (the lowest value will be recorded)
Percentage of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | From baseline by visit up to week 28 (study visit 9, Follow-Up)
  Clinically significant changes in ECGs from baseline by visit. ECGs should be collected in triplicate, 1 to 3 minutes apart, and read locally
Percentage of patients with clinically significant changes in physical examination | From baseline by visit up to week 28 (study visit 9, Follow-Up)
  Clinically significant changes in physical examinations from baseline by visit. Physical examinations will include general appearance, skin, head, ears, eyes, nose, throat, neck, lungs, heart, abdomen, musculoskeletal, extremities, and neurological systems
Percentage of patients with clinically significant changes in hematology, serum chemistry, urinalysis, and thyroid function | From baseline by visit up to week 28 (study visit 9, Follow-Up)
  Clinically significant changes in hematology, serum chemistry, urinalysis, and thyroid function from baseline by visit
Percentage of patients with clinically significant changes in hearing audiometric testing (bone- and air-conduction) | From baseline by visit up to week 28 (study visit 9, Follow-Up)
  Clinically significant changes in hearing audiometric testing from baseline by visit. Pure tone audiometry (PTA) air conduction thresholds will be conducted at frequencies 250, 500, 1000, 2000, 4000, and 8000 Hz. Bone conduction thresholds will be conducted at frequencies 500, 1000, 2000, and 4000 Hz.

CONTACTS AND LOCATIONS:
Locations (17):
- Medizinische Universitaet Wien, Vienna, Vienna, Austria
- Czechia (4):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - Institut Klinicke a Experimentalni Mediciny, Prague
  - Vseobecna Fakultni Nemocnice v Praze, Prague
- AP-HP Hopital Necker-Enfants Malades, Paris, France
- Spain (7):
  - Hospital Universitario 12 de Octubre, Madrid, Usera
  - Fundacio Puigvert, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Fundacion Jimenez Diaz, Madrid
- United Kingdom (4):
  - Royal Free London NHS Foundation Trust, London
  - Great Ormond Street Hospital for Children, London
  - Royal Manchester Children's Hospital, Manchester
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rheault MN. Treatment Approaches for Alport Syndrome. J Am Soc Nephrol. 2025 Sep 12;37(1):172-9. doi: 10.1681/ASN.0000000897. Online ahead of print. PMID 40938675